CLINICAL TRIAL: NCT00901524
Title: ANRS HC20 Pilot Study, Multicenter, Assessing the Effectiveness of an Optimized Anti HCV (360μg/Week Induction of PegIFN-alpha2a + 18mg/kg/j of RBV for 6 Months and Then Depending on the Virological Response to S12, Elongation up S72 to the Dual Anti HCV, With Accompanying Measures) on Sustained Virological Response in Patients With HCV Genotype 1 and 4 Non Responders and Co-infected With HIV.
Brief Title: ANRS HC20 Effectiveness of an Optimized Anti HCV PegIFN-alpha2a + Ribavirin on Sustained Virological Response in Patients With HCV Genotype 1 and 4 Non Responders and Co-infected With HIV
Acronym: ETOC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008-000859-10; ANRS HC 20
Record Dates: First submitted 2009-04-28; First posted 2009-05-13 (Estimated); Last update posted 2013-03-29 (Estimated); Status verified 2012-10

CONDITIONS: Hepatitis
Keywords: HCV Genotype 1, 4; Virological response; Ribavirin; PegPegIFN- alpha 2a; Viral Hepatitis (HCV)
MeSH Terms: conditions — Hepatitis; Hepatitis C | interventions — Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PegIFN- alpha 2a + RBV (No Intervention)
  Interventions: Drug: Peg-interféron alpha 2a + ribavirin

INTERVENTIONS:
Drug: Peg-interféron alpha 2a + ribavirin — Pilot study, multicenter, open label

SUMMARY:
The purpose of this study is to assess the effectiveness of an optimized anti HCV treatment (360μg per week of PegIFN-alpha2a + 18mg/kg/j of Ribavirin for 6 months.

DETAILED DESCRIPTION:
In patients HIV infected, the success rate do not exceed 20% in genotype 1 or 4 patients. In case of treatment failure , patients are rarely re-treated, and liver fibrosis progresses rapidly. The new molecules are not yet available for patients co-infected with HIV, and patients having already undergone a first treatment will likely be among the last to be included in trials evaluating the effectiveness of these treatments.

However, recent studies show that it is possible to propose a new treatment "optimized" to these patients in the hope to obtain better success rate. Provide antiretroviral treatment, use of high doses of Peg-interferon and ribavrine, and supporting patients.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Weight 85 kg below the pre-inclusion visit.
* Documented HIV infection (HIV positive)
* HCV infection documented by a positive PCR
* HCV Genotype 1 or 4
* Compensated liver disease (Child-Pugh below/equal to 6)
* Lymphocytes CD4 above 200/mm3
* Patient not answering a treatment for hepatitis C.
* Patient not covered by dual by Peg-IFN + riba for at least three months (wash out)

Exclusion Criteria:

* Co-infection with HBV (HBsAg positive)
* Neutropenia below 1000/mm3
* Thrombocytopenia below 90000/mm3 or thrombocytosis over 500 000/mm3.
* Hemoglobin below 11 g / dL (men and women)
* Arguments radiological (ultrasound, CT or MRI) of hepatocellular carcinoma cell
* Antiretroviral containing didanosine (ddI) and stavudine (d4T) and zidovudine (AZT) and abacavir (ABC).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2009-06; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Study the proportion of patients co-infected HIV-HCV, non-responders to treatment for HCV (genotype 1 and 4), with a sustained virological response (6 months after stopping treatment (W72 or W96)) at a re-optimized treatment of hepatitis C. | W72 or W96 (depending of the end of treatment)

SECONDARY OUTCOMES:
Analyze rapid virological response (W4) and early (W12). | W4 and W12

CONTACTS AND LOCATIONS:
Overall Officials: Philippe BONNARD, MD, Principal Investigator — Hopital Tenon
Locations (1):
- Hôpital Tenon Service des Maladies Infectieuses, Paris, France

REFERENCES:
- [Derived] Laird ME, Mohsen A, Duffy D, Mamdouh R, LeFouler L, Casrouge A, El-Daly M, Rafik M, Abdel-Hamid M, Soulier A, Pawlotsky JM, Hezode C, Rosa I, Renard P, Mohamed MK, Bonnard P, Izopet J, Mallet V, Pol S, Albert ML, Fontanet A. Apolipoprotein H expression is associated with IL28B genotype and viral clearance in hepatitis C virus infection. J Hepatol. 2014 Oct;61(4):770-6. doi: 10.1016/j.jhep.2014.05.040. Epub 2014 Jun 4. PMID 24905490
- See also: French National Agency for Research on AIDS and Viral Hepatitis website — http://www.anrs.fr